CLINICAL TRIAL: NCT03644368
Title: Retrospective Evaluation of the Management of Children's Deep Neck Infections at the Montpellier Hospital
Brief Title: Children's Deep Neck Infections at the Montpellier Hospital
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0212
Record Dates: First submitted 2018-07-02; First posted 2018-08-23 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-07

CONDITIONS: Deep Neck Infections
Keywords: cervical phlegmon; tonsillar abscesses; retropharyngeal or parapharyngeal abscesses; medical and chirurgical treatment; Bacteria in deep neck infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To descride the clinical presentation, diagnosis, management and complications of children with a deep neck infection. A retrospective chart review was conducted at the Montpellier hospital in France. All children aged less than 18 years who had been admitted with a diagnosis of cervical phlegmon, tonsillar abscesses, retropharyngeal or parapharyngeal abscesses between January 2015 and December 2017 were included. The investigators collected the demographic, biological, radiological data and treatment received of the patients to the admision. The results of the bacteriological samples were collected. The investigators compared our results to those of the 10-year cohort. The investigators wish to compare the duration of hospitalization and the duration of the fever enter the group treated by alone antibiotic and the group treated by antibiotic and surgical drainage

ELIGIBILITY:
Inclusion criteria:

* under 18 years old
* hospitalized for acute pharyngeal infection ( cervical phlegmon, tonsillar abscesses, retropharyngeal or parapharyngeal abscesses)

Exclusion criteria:

* neck infection in the context of immune deficiency
* malignancy or post-traumatic disease
* others deep neck infections: angina, otitis, sinusitis, ethmoiditis, mastoiditis.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children hospitalized for acute pharyngeal infection
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Clinical description of acute peripharyngeal suppuration | 1 day
  Clinical description of acute peripharyngeal suppuration suppuration

SECONDARY OUTCOMES:
Description of therapeutic management | 1 day
  Description of therapeutic management : vaccinations, treatments received before hospitalization, treatments received during hospitalization
Description of bacteria in deep neck infections | 1 day
  Description of bacteria in deep neck infections

OTHER OUTCOMES:
duration of hospitalization | 1 day
  Compare the duration of hospitalization enter the group treated by alone antibiotic and the group treated by antibiotic and surgical drainage.
duration of the fever | 1 day
  Compare the duration of the fever enter the group treated by alone antibiotic and the group treated by antibiotic and surgical drainage.

CONTACTS AND LOCATIONS:
Overall Officials: Eric JEZIORSKI, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC